CLINICAL TRIAL: NCT05369143
Title: The Effects of Chiropractic Care on Neurophysiological Function Immune Markers and Health Related Quality of Life in Children With Subclinical Spinal Pain Using Artificial Intelligence Modelling
Brief Title: The Effects of Chiropractic Care and Children With Subclinical Spinal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/01286 Imran Amjad
Record Dates: First submitted 2022-04-26; First posted 2022-05-11 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Subclinical Spinal Pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiropractic care Group (Experimental): A registered chiropractor will assess the entire spine, and both sacroiliac joints will be assessed for vertebral subluxation by a registered chiropractor with at least five years of clinical experience.The clinical indicators that will be used to assess the function of the spine before spinal adjustment intervention include assessing for joint tenderness to palpation manually palpating for a restricted intersegmental range of motion, assessing for palpable asymmetric intervertebral muscle tension, and any abnormal or blocked joint play and end-feel of the joints. Chiropractors use these biomechanical characteristics as clinical indicators of spinal dysfunction and vertebral subluxation.
  Interventions: Other: Chiropractic care
- Control Group (Placebo Comparator): The participants head and/or spine will be moved in ways that include passive and active movements, similar to what is done when assessing the spine by a chiropractor. The control intervention will also include the participants moving into adjustment setup positions similar to how the chiropractor would typically set up a patient with no joint pre-loading or adjustive thrust. No spinal adjustment will be performed during any control intervention. This control intervention is not intended to act as a sham treatment session
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Chiropractic care — The mechanical properties of chiropractic adjustment have been investigated; and although the actual force applied to the patient's spine depends on the chiropractor, the patient, and the spinal location of the subluxation, the general shape of the force-time history of spinal adjustments is very consistent68 and the duration of the thrust is always less than 200 milliseconds.
  Arms: Chiropractic care Group
Other: Control Group — The participants head and/or spine will be moved in ways that include passive and active movements, similar to what is done when assessing the spine by a chiropractor. The sham intervention will also include the participants moving into adjustment setup positions similar to how the chiropractor would typically set up a patient with no joint pre-loading or adjustive thrust
  Arms: Control Group

SUMMARY:
There is growing evidence that chiropractic care positively impacts various aspects of central and autonomic nervous system function.This study aims to investigate short term and long-term effects of Chiropractic care (CC) on neurological, behavioral, immunological functions and health-related quality of life in children with subclinical spinal pain.

DETAILED DESCRIPTION:
There is growing evidence that chiropractic care positively impacts various aspects of central and autonomic nervous system function. A single chiropractic adjustment session has been shown to alter pre-frontal cortex (PFC) activity in adults, but there is a lack of robust research investigating any long-term benefits of such PFC changes in children. This study aims to investigate short term and long-term effects of Chiropractic care (CC) on neurological, behavioral, immunological functions and health-related quality of life in children with subclinical spinal pain. In this parallel-group randomized controlled trial, participants aged 10-18 years with subclinical spinal pain will be randomly allocated to receive either 12 weeks of CC intervention or control intervention. Primary outcomes include functional near-infrared spectroscopy, heart rate variability (HRV) and resting-state electroencephalography (EEG). The secondary outcomes include executive functions measured by cognitive testing, immune and inflammation status, and health-related quality of life. As data collected in the project is the combination of extrinsic (sociodemographic, clinical questionnaires etc.) and intrinsic physiological data (physiological measures like EEG, HRV etc.), we will utilize the advances in machine learning or artificial intelligence (AI) to help inform the development of optimal chiropractic care plans in future.

ELIGIBILITY:
Inclusion Criteria:

* aged between 10 and 18 years
* have subclinical spinal pain

Exclusion Criteria:

* no evidence of spinal dysfunction is present
* they are in current pain (above 3/10 on VAS)
* have sought previous treatment for their spinal issues
* are unable to perform the assessment procedures due to contraindications or movement limitations
* diagnosed immune dysfunction
* utilizing a prescribed immunosuppressive medication
* have uncontrolled asthma
* nasal polyps
* use of an intranasal steroid spray one month or less before the study
* are HIV-positive
* are participating in another research study at the time of data collection
* have any diagnosed comorbidity or concomitant disease
* have allergies to yeast or yeast-derived products
* have chronic sinusitis or recent (within the last six weeks) episode of acute sinusitis.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Functional near-infrared spectroscopy (fNIRS) | Base line
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks (Cognitive tasks). A baseline assessment of a participant will be done before the start of the intervention.
Functional near-infrared spectroscopy (fNIRS) | After 6 weeks of intervention
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks (Cognitive tasks). Assessment of participants will be repeated after 6 weeks of intervention.
Functional near-infrared spectroscopy (fNIRS) | After 12 weeks of intervention and 16 weeks (4-week follow-up testing in a sub-group of participants. )
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks (Cognitive tasks). Assessment of participants will be repeated after 12 weeks of intervention.
Functional near-infrared spectroscopy (fNIRS) | After 16 weeks of intervention
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks (Cognitive tasks). Assessment of participants will be repeated after 16 weeks of intervention.
Heart rate variability | Up to 16 Weeks
  Heart rate variability (HRV) will be used as an objective assessment of psychological health and stress for the participants. High HRV is a marker of an adaptable, responsive nervous system that can detect sensory stimuli and appropriately increase or decrease the heart rate based on the needs of the individual. Low HRV and low parasympathetic activity is associated with chronic pain states, poor cardiovascular health and mood disorders. Heart Rate will be monitored throughout the session. Assessment of participants will be continued throughout the intervention.
Whole head EEG(sub-cohort of participants) | Base line
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention.
  A baseline assessment will be done before applying intervention.
Whole head EEG(sub-cohort of participants) | After 6 weeks of intervention
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention. Assessment of participants will be repeated after 6 weeks of intervention.
Whole head EEG(sub-cohort of participants) | After 12 weeks of intervention
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention. Assessment of participants will be repeated after 12 weeks of intervention.
Whole head EEG(sub-cohort of participants) | After 16 weeks of intervention
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention. Assessment of participants will be repeated after 16 weeks of intervention.

SECONDARY OUTCOMES:
Spatial working memory (SWM) | Base line
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has notable executive function demands and provides a measure of strategy as well as working memory error.
  Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes that have already been found to contain a token) and strategy.
  Fewer errors mean good spatial working memory and vice versa for more errors. A baseline assessment of a participant will be done before the start of the intervention.
Spatial working memory (SWM) | After 6 weeks of intervention
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has notable executive function demands and provides a measure of strategy as well as working memory error.
  Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes that have already been found to contain a token) and strategy.
  Fewer errors mean good spatial working memory and vice versa for more errors. Assessment of participants will be repeated after 6 weeks of intervention.
Spatial working memory (SWM) | After 12 weeks of intervention
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has notable executive function demands and provides a measure of strategy as well as working memory error.
  Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes that have already been found to contain a token) and strategy.
  Fewer errors mean good spatial working memory and vice versa for more errors. Assessment of participants will be repeated after 12 weeks of intervention.
Spatial working memory (SWM) | After 16 weeks of intervention
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has notable executive function demands and provides a measure of strategy as well as working memory error.
  Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes that have already been found to contain a token) and strategy.
  Fewer errors mean good spatial working memory and vice versa for more errors. Assessment of participants will be repeated after 16 weeks of intervention.
Reaction time (RTI) | Base line
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  It's a six-minute test that covers latency (response speed), correct responses and errors of commission and omission.
  More accurate reaction in less time inclines toward good reaction time. A baseline assessment of a participant will be done before the start of the intervention.
Reaction time (RTI) | After 6 weeks of intervention
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  It's a six-minute test that covers latency (response speed), correct responses and errors of commission and omission.
  More accurate reaction in less time inclines toward good reaction time. Assessment of participants will be repeated after 6 weeks of intervention.
Reaction time (RTI) | After 12 weeks of intervention
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  It's a six-minute test that covers latency (response speed), correct responses and errors of commission and omission.
  More accurate reaction in less time inclines toward good reaction time. Assessment of participants will be repeated after 12 weeks of intervention.
Reaction time (RTI) | After 16 weeks of intervention
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  It's a six-minute test that covers latency (response speed), correct responses and errors of commission and omission.
  More accurate reaction in less time inclines toward good reaction time. Assessment of participants will be repeated after 16 weeks of intervention.
Paired Associate Learning (PAL) | Base line
  Paired Associates Learning assesses visual memory and new learning Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed. A baseline assessment of a participant will be done before the start of the intervention.
Paired Associate Learning (PAL) | After 6 weeks of intervention
  Paired Associates Learning assesses visual memory and new learning Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed. Assessment of participants will be repeated after 6 weeks of intervention.
Paired Associate Learning (PAL) | After 12 weeks of intervention
  Paired Associates Learning assesses visual memory and new learning Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed. Assessment of participants will be repeated after 12 weeks of intervention.
Paired Associate Learning (PAL) | After 16 weeks of intervention
  Paired Associates Learning assesses visual memory and new learning Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed. Assessment of participants will be repeated after 16 weeks of intervention.
Stockings of Cambridge (SoC) | At Baseline
  Stockings of Cambridge (SOC) is a test of spatial planning that requires individuals to use problem-solving strategies to match two sets of stimuli. A baseline assessment of a participant will be done before the start of the intervention.
Stockings of Cambridge (SoC) | After 6 weeks of intervention
  Stockings of Cambridge (SOC) is a test of spatial planning that requires individuals to use problem-solving strategies to match two sets of stimuli.
  Assessment of participants will be repeated after 6 weeks of intervention.
Stockings of Cambridge (SoC) | After 12 weeks of intervention
  Stockings of Cambridge (SOC) is a test of spatial planning that requires individuals to use problem-solving strategies to match two sets of stimuli. Assessment of participants will be repeated after 12 weeks of intervention.
Stockings of Cambridge (SoC) | After 16 weeks of intervention
  Stockings of Cambridge (SOC) is a test of spatial planning that requires individuals to use problem-solving strategies to match two sets of stimuli. Assessment of participants will be repeated after 16 weeks of intervention.
Delayed Matching to Sample (DMS) | At Baseline
  Delayed Matching to Sample assesses both simultaneous visual matching ability and short-term visual recognition memory for non-verbalizable patterns. A baseline assessment of a participant will be done before the start of the intervention.
Delayed Matching to Sample (DMS) | After 6 weeks of intervention
  Delayed Matching to Sample assesses both simultaneous visual matching ability and short-term visual recognition memory for non-verbalizable patterns. Assessment of participants will be repeated after 6 weeks of intervention.
Delayed Matching to Sample (DMS) | After 12 weeks of intervention
  Delayed Matching to Sample assesses both simultaneous visual matching ability and short-term visual recognition memory for non-verbalizable patterns. Assessment of participants will be repeated after 12 weeks of intervention.
Delayed Matching to Sample (DMS) | After 16 weeks of intervention
  Delayed Matching to Sample assesses both simultaneous visual matching ability and short-term visual recognition memory for non-verbalizable patterns. Assessment of participants will be repeated after 16 weeks of intervention.
Health-related quality of life | Base line
  The health-related quality of life will be measured using the PROMIS Pediatric v2.0 profile 25, which assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. PROMIS Pediatric v2.0 profile 25 is a reliable and valid instrument that can be used to assess the impacts of health care interventions and track changes in health over time. A baseline assessment of a participant will be done before the start of the intervention.
  The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112.
Health-related quality of life | After 6 weeks of intervention
  The health-related quality of life will be measured using the PROMIS Pediatric v2.0 profile 25, which assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. PROMIS Pediatric v2.0 profile 25 is a reliable and valid instrument that can be used to assess the impacts of health care interventions and track changes in health over time. Assessment of participants will be repeated after 6 weeks of intervention.
  The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112.
Health-related quality of life | After 12 weeks of intervention
  The health-related quality of life will be measured using the PROMIS Pediatric v2.0 profile 25, which assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. PROMIS Pediatric v2.0 profile 25 is a reliable and valid instrument that can be used to assess the impacts of health care interventions and track changes in health over time. Assessment of participants will be repeated after 12 weeks of intervention.
  The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112.
Health-related quality of life | After 16 weeks of intervention
  The health-related quality of life will be measured using the PROMIS Pediatric v2.0 profile 25, which assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. PROMIS Pediatric v2.0 profile 25 is a reliable and valid instrument that can be used to assess the impacts of health care interventions and track changes in health over time. Assessment of participants will be repeated after 16 weeks of intervention.
  The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112.

OTHER OUTCOMES:
Saliva Cortisol | Base line
  Cortisol can alter cytokine levels (such as increasing IL-6 pro-inflammatory cytokines) that then alter the levels of inflammation throughout the body. Cortisol could be measured from saliva samples.
  Cortisol (otherwise known as the stress hormone) is made in the adrenal glands. It's elevated when we experience heightened anxiety or stress, and it's lowered when we're in a relaxed state. A baseline assessment of a participant will be done before the start of the intervention.
Saliva Cortisol | after 12 weeks of intervention
  Cortisol can alter cytokine levels (such as increasing IL-6 pro-inflammatory cytokines) that then alter the levels of inflammation throughout the body. Cortisol could be measured from saliva samples.
  Cortisol (otherwise known as the stress hormone) is made in the adrenal glands. It's elevated when we experience heightened anxiety or stress, and it's lowered when we're in a relaxed state. Assessment of participants will be repeated after 12 weeks of intervention.
Saliva Cortisol | after 16 weeks of intervention
  Cortisol can alter cytokine levels (such as increasing IL-6 pro-inflammatory cytokines) that then alter the levels of inflammation throughout the body. Cortisol could be measured from saliva samples.
  Cortisol (otherwise known as the stress hormone) is made in the adrenal glands. It's elevated when we experience heightened anxiety or stress, and it's lowered when we're in a relaxed state. Assessment of participants will be repeated after 16 weeks of intervention.
Hair Cortisol | Baseline
  Cortisol can alter cytokine levels (such as increasing IL-6 pro-inflammatory cytokines) that then alter the levels of inflammation throughout the body. Cortisol could be measured from Hair samples.
  Cortisol (otherwise known as the stress hormone) is made in the adrenal glands. It's elevated when we experience heightened anxiety or stress, and it's lowered when we're in a relaxed state. Assessment of participants will be done at the baseline of the study.
Hair Cortisol | After 12 weeks of intervention
  Cortisol can alter cytokine levels (such as increasing IL-6 pro-inflammatory cytokines) that then alter the levels of inflammation throughout the body. Cortisol could be measured from Hair samples.
  Cortisol (otherwise known as the stress hormone) is made in the adrenal glands. It's elevated when we experience heightened anxiety or stress, and it's lowered when we're in a relaxed state. Assessment of participants will be repeated after 12 weeks of intervention.
Immune Function Questionnaire (IFQ) | At baseline
  The Immune Function Questionnaire (IFQ) consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and prolonged healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. A baseline assessment of a participant will be done before the start of the intervention.
  Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status.
Immune Function Questionnaire (IFQ) | After 6 weeks of intervention
  The Immune Function Questionnaire (IFQ) consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and prolonged healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be repeated after 6 weeks of intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status.
Immune Function Questionnaire (IFQ) | After 12 weeks of intervention
  The Immune Function Questionnaire (IFQ) consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and prolonged healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be repeated after 12 weeks of intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status.
Immune Function Questionnaire (IFQ) | After 16 weeks of intervention
  The Immune Function Questionnaire (IFQ) consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and prolonged healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be repeated after 16 weeks of intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status.
Inflammation markers from Fitbit data | Up to 16 Weeks
  Fitbit can be used to measure the autonomic nervous system (ANS). Heart rate variability (HRV) has become a validated marker of autonomic function. In a large population-based study it was found that strong and independent relationships between HR and HRV with a broad set of inflammatory biomarkers. The recording will be done for up to 16 weeks.
Smartphone Gait and Balance Application | Baseline
  The system consists of the following three components: i) a smartphone that has an embedded accelerometer, ii) a belt to house the phone on the lower back, iii) and a smartphone balance application. There are six different tasks that the subject has to perform with the system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and closed and standing on a compromised surface with eyes open and closed. This app. will calculate mediolateral and anterior-posterior sway during each task. Assessment will be done at baseline.
Smartphone Gait and Balance Application | After 6 weeks of intervention
  The system consists of the following three components: i) a smartphone that has an embedded accelerometer, ii) a belt to house the phone on the lower back, iii) and a smartphone balance application. There are six different tasks that the subject has to perform with the system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and closed and standing on a compromised surface with eyes open and closed. This app. will calculate mediolateral and anterior-posterior sway during each task. Assessment will be done after 6 weeks.
Smartphone Gait and Balance Application | After 12 weeks of intervention
  The system consists of the following three components: i) a smartphone that has an embedded accelerometer, ii) a belt to house the phone on the lower back, iii) and a smartphone balance application. There are six different tasks that the subject has to perform with the system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and closed and standing on a compromised surface with eyes open and closed. This app. will calculate mediolateral and anterior-posterior sway during each task. Assessment will be done after 12 weeks.
Smartphone Gait and Balance Application | After 16 weeks of intervention
  The system consists of the following three components: i) a smartphone that has an embedded accelerometer, ii) a belt to house the phone on the lower back, iii) and a smartphone balance application. There are six different tasks that the subject has to perform with the system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and closed and standing on a compromised surface with eyes open and closed. This app. will calculate mediolateral and anterior-posterior sway during each task. Assessment will be done after 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: IMRAN KHAN NIAZI, PhD, Principal Investigator — New Zealand College of Chiropractic
Locations (1):
- Mera Ghar Orphan House, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No